CLINICAL TRIAL: NCT03560011
Title: Efficacy and Safety of Immunoglobulin Associated With Rituximab Versus Rituximab Alone in Childhood-Onset Steroid-dependent Nephrotic Syndrome
Acronym: RITUXIVIG
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Decision of Data Safety Monitoring Board
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160905J; 2017-000826-36 (EudraCT Number)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Steroid-Dependent Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — gamma-Globulins

STUDY DESIGN:
Intervention Model Description: 2 Arms :
  * Rituximab (375 mg/m2)
  * Rituximab (375 mg/m2) followed by 5 injections of immunoglobulin IV once a month during 5 months (2g/kg at M1, 1.5g/kg at M2 to M5, maximal dise 100g)
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (375 mg/m²) (No Intervention): Single infusion of rituximab (375 mg/m²)
- Rituximab followed by 5 injections of immunoglobulin IV (Experimental): Rituximab (375 mg/m²) followed by 5 injections of immunoglobulin IV once a month during 5 months (2g/kg at M1, 1.5g/kg at M2 to M5, maximal dose 100g). Treatment duration : 6 months
  Interventions: Drug: immunoglobulin IV

INTERVENTIONS:
Drug: immunoglobulin IV — 5 injections of immunoglobulin IV once a month during 5 months (2g/kg at M1, 1.5g/kg at M2 to M5, maximal dose 100g)
  Arms: Rituximab followed by 5 injections of immunoglobulin IV

SUMMARY:
Idiopathic Nephrotic Syndrome (INS) is the first glomerulopathy in children and 60% of the patients develop Steroid-Dependant Nephrotic Syndrome (SDNS). Recently, rituximab (RTX), a humanized anti-CD20 antibody depleting B cells demonstrated the ability to increase relapse free survival and to decrease the number of relapse and the need of other immunosuppressive drugs. However, the remission rate after 2 years is only 30 to 40%.

The aim of the study is to study the ability of intravenous Immunoglobulin to improve remission rate in SDNS when added associated with Rituximab compared to a treatment by Rituximab alone.

DETAILED DESCRIPTION:
Idiopathic Nephrotic Syndrome (INS) is the first glomerulopathy in children and 60% of the patients develop Steroid-Dependant Nephrotic Syndrome (SDNS). Depleting B cells demonstrated the ability to increase relapse free survival and to decrease the number of relapse and the need of other immunosuppressive drugs. However, the remission rate after 2 years is only 30 to 40%.

The aim of the study is to study the ability of intravenous Immunoglobulin to improve remission rate in SDNS when added associated with Rituximab compared to a treatment by Rituximab alone.

ELIGIBILITY:
Inclusion Criteria:

* Childhood onset nephrotic syndrome (first flair <18 years)
* ≥ 2 years old at inclusion
* Steroid-dependent:

  * Patient with at least 2 relapses confirmed during the decay of corticosteroids or within 2 weeks following steroids discontinuation.
  * Patient with at least 2 relapses including one under steroidsparing agent (MMF, Calcineurin inhibitors, cyclophosphamide, Levamisole) or within 6 months of treatment withdrawal.
* or with frequent relapses:

  · 2 or more relapses within 6 months after initial remission or 4 or more relapses within any 12-month period.
* with a relapse within 3 months prior to inclusion
* In remission: Protein-over-creatinine ratio ≤ 0.2g/g (≤ 0.02g/mmol)

Exclusion Criteria:

* Patients with steroid-resistant nephrotic syndrome;
* Patients with genetic nephrotic syndrome;
* Patients previously treated with rituximab;
* Patients with no affiliation to a social security scheme (beneficiary or legal);
* Prior Hepatitis B, Hepatitis C or HIV infection;
* Pregnancy or breastfeeding.
* Patients with hyperprolinaemia,
* Known hypersensitivity to one of the study medication,
* Scheduled and not postponable injection of live attenuated vaccine
* Protected adults
* Patients with neutrophils < 1.5 G/L and/or platelets < 75 G/L

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2022-11-04 (Estimated)

PRIMARY OUTCOMES:
The occurrence of the first relapse | 24 months
  Relapse is defined as a protein to creatinine ratio of 2g/g of creatinine (0.2 g/mmol) or higher

SECONDARY OUTCOMES:
Time to first relapse | 24 months
Number of relapse over a 24 months follow-up | 24 months
Cumulative amount of corticosteroid over a 24 months follow-up | 24 months
Adverse events in each arm | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien HOGAN, MD PhD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526
- [Derived] Chan EY, Yap DY, Colucci M, Ma AL, Parekh RS, Tullus K. Use of Rituximab in Childhood Idiopathic Nephrotic Syndrome. Clin J Am Soc Nephrol. 2023 Apr 1;18(4):533-548. doi: 10.2215/CJN.08570722. Epub 2023 Feb 22. PMID 36456193
- [Derived] Hogan J, Perez A, Sellier-Leclerc AL, Vrillon I, Broux F, Nobili F, Harambat J, Bessenay L, Audard V, Faudeux C, Morin D, Pietrement C, Tellier S, Djeddi D, Eckart P, Lahoche A, Roussey-Kesler G, Ulinski T, Boyer O, Plaisier E, Cloarec S, Jolivot A, Guigonis V, Guilmin-Crepon S, Baudouin V, Dossier C, Deschenes G. Efficacy and safety of intravenous immunoglobulin with rituximab versus rituximab alone in childhood-onset steroid-dependent and frequently relapsing nephrotic syndrome: protocol for a multicentre randomised controlled trial. BMJ Open. 2020 Sep 23;10(9):e037306. doi: 10.1136/bmjopen-2020-037306. PMID 32967877